CLINICAL TRIAL: NCT04535973
Title: Hormonal Status and Quality of Life in Female Postmenopausal Patients With Burning Mouth Syndrome
Status: Completed | Type: Observational
Sponsor: University of Zagreb (Other)
Responsible Party: Principal Investigator, Božana Lončar Brzak, Assistant Professor, University of Zagreb
Other Study IDs: Univ Zg
Record Dates: First submitted 2020-08-22; First posted 2020-09-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Burning Mouth Syndrome; Progesterone; Dehydroepiandrosterone; Quality of Life; Hormone Disturbance; 17β-Estradiol
Keywords: burning mouth syndrome; hormonal status; quality of life
MeSH Terms: conditions — Burning Mouth Syndrome; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: female postmenopausal women with burning mouth syndrome
  Interventions: Diagnostic Test: unstimulated saliva sample for hormone analysis; Other: quality of life questionnaire
- control group: female postmenopausal women without burning mouth syndrome
  Interventions: Diagnostic Test: unstimulated saliva sample for hormone analysis; Other: quality of life questionnaire

INTERVENTIONS:
Diagnostic Test: unstimulated saliva sample for hormone analysis — hormone levels will be determined in frozen samples of unstimulated saliva
Other: quality of life questionnaire — all participants will fill out self-perceived quality of life questionnaire

SUMMARY:
The aim of this study was to determine the level of salivary estradiol, progesterone and dehydroepiandrosterone in female postmenopausal women with and without burning mouth syndrome. In all participants the quantity of unstimulated and stimulated saliva would be determined and they would fulfill self-perceived quality of life questionnaire Oral Health Impact Profile-14 (OHIP-14). Intensity of burning symptoms would be determined on visual-analogue scale grading 0-10. All data would be compared between study and control group.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal women with burning mouth syndrome

Exclusion Criteria:

* women with burning mouth syndrome who are not in menopause

Ages: 51 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Study Population: postmenopausal women are most frequently affected with burning mouth syndrome, and we wanted the groups to be as similar as possible so we included only postmenopausal women, with and without burning mouth syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
to evaluate the levels of salivary hormone | November 2019-June 2020
  levels of salivary 17β-Estradiol, progesterone and DHEA were determined in study and control group

SECONDARY OUTCOMES:
to evaluate quality of life and correlate it with levels of salivary hormones and intensity of symptoms | November 2019-June 2020
  quality of life was evaluated with self-perceived questionnaire OHIP-14

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dental Medicine, University of Zagreb, Zagreb, Croatia